CLINICAL TRIAL: NCT05419765
Title: Nonalcoholic Fatty Liver Disease: Crosstalk Between Genetic Predisposition and Epigenetic Lysosomal Acid Lipase Activity Reduction in Blood, Plasma and Platelets
Brief Title: Lysosomal Acid Lipase Activity in Nonalcoholic Fatty Liver Disease
Acronym: NAFLD LAL
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, STEFANO GINANNI CORRADINI, Associate Professor, University of Roma La Sapienza
Other Study IDs: Sapienza Univ&Alexion Pharma
Record Dates: First submitted 2022-05-26; First posted 2022-06-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2022-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Lysosomal acide lipase; PNPLA3; TM6SF2; HSD17B13; Hepatic elastography
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- non-cirrhotic NAFLD, carriers of the PNPLA3 I148M variant: Italian Caucasians, aged> 18 and <70 years, with non-cirrhotic NAFLD and carriers of the PNPLA3 I148M variant
  Interventions: Diagnostic Test: Peripheral blood withdrawn
- non-cirrhotic NAFLD, carriers of the wild type allele: Italian Caucasian subjects, aged> 18 and <70 years, with non-cirrhotic NAFLD and carriers of the wild type allele
  Interventions: Diagnostic Test: Peripheral blood withdrawn

INTERVENTIONS:
Diagnostic Test: Peripheral blood withdrawn — Peripheral blood will be withdrawn in order to measure haematic lipids (total cholesterol and fractions, triglycerides), total blood LAL activity, to perform genetic analysis and finally to evaluate lipase activity into the platelets.
  Hepatic elastography will be also executed, in 100 patients, according to the presence/absence of the PNPLA3 variant, in order to weigh up the genetic predisposition on NAFLD development or progression
  Other Names: Hepatic elastography

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a multifactorial disease affecting a quarter of the world population. Pathological accumulation of fat, into the hepatocytes, is the first hit and is due to altered hepatic and extrahepatic lipogenesis, lipolysis and lipophagy of the large lipid droplets.

Lipophagy plays a key role in the onset of NAFLD, in the autolysosomes, small droplets of fat are catabolized by Lysosomal Acid Lipase (LAL) enzyme which hydrolyzes cholesterol esters and triglycerides forming cholesterol and free fatty acids.

Our research group demonstrated that, subjects affected by NAFLD, present a reduced enzymatic activity either compared to patients with chronic liver disease of different etiology, but comparable staging, either compared to healthy control subjects.

Leukocytes are the main site of enzymatic activity in the blood, however, our research group has shown that it can also be detected inside the platelets, demonstrating how the LAL activity can be exchanged between cells.

Furthermore, our group has shown, for the first time, how the intracellular enzymatic activity is reduced, independently of the platelets and leukocytes count and progressively from chronic liver disease up to cirrhosis.

Among factors which contribute to altered lipid metabolism, the genetic predisposition to the accumulation of hepatic fat must be counted. Several variants of genes that code for proteins implicated in the digestion or storage of fats, are involved.

In this study were considered: patatin-like phospholipase domain-containing 3 (PNPLA3), Transmembrane 6 superfamily 2 (TM6SF2) and 17β-Hydroxysteroid dehydrogenase type 13 (HSD17B13).

The rs738409 variant (C> G, p.I148M) of the PNPLA3 gene consists of a protein in which the catalytic site is not entirely accessible to the substrate which, consequently, accumulates in the storage site.

This variant is commonly found in NAFLD subjects and it has been widely reported how the variant carriers progress faster towards severe disease (steatohepatitis) than wild type subjects.

The TM6SF2 gene encodes a membrane transporter involved in the triglycerides movement, the rs58542926 (C> T E167K) variant has been associated with an increased predisposition towards liver fibrosis in NAFLD subjects. This is likely due to the loss of protein function resulting in hepatic retention of triglycerides and cholesterol.

Unlike PNPLA3 and TM6SF2, the rs72613567 (TA> TAA) variant of the HSD17B13 gene has a protective effect against NAFLD progression. It is characterized by a protein loss of function that protects against chronic liver damage and mitigates the progression of the disease although how the protective effect occurs is still under study.

Due to the multifactorial etiology of the disease, to the need of carrying out a targeted surveillance in predisposed genetic subjects and, in order to prevent NALFD progression towards severe pathological forms characterized by an increased mortality, in this study, 316 subjects will be enrolled.

They will be divided as follows: Italian Caucasians, aged> 18 and <70 years, with non-cirrhotic NAFLD and carriers of the PNPLA3 I148M variant, and, 158 Italian Caucasian subjects, aged> 18 and <70 years, with non-cirrhotic NAFLD and carriers of the wild type allele.

The following exclusion criteria will be considered: any type of malignant disease in the past 5 years, any type of inflammatory or autoimmune disease, corticosteroids for systemic use, any type of drug that may affect body weight or body composition, insufficiency kidney (GFR <90 mL / min), heart failure (NYHA classes II-IV), any type of liver disease rather than NAFLD, excessive alcohol intake (> 140 g / week for men and 70 g / week for women), participation in a weight reduction program in the past 3 months, bile salts, cholestyramine in the last 6 months prior to enrollment, previous cholecystectomy, gallbladder disease.

Peripheral blood will be withdrawn in order to measure haematic lipids (total cholesterol and fractions, triglycerides), total blood LAL activity, to perform genetic analysis and finally to evaluate lipase activity into the platelets.

Hepatic elastography will be also executed, in 100 patients, according to the presence/absence of the PNPLA3 variant, in order to weigh up the genetic predisposition on NAFLD development or progression Finally, in subjects who present a lipase activity 30% lower than the normal value (0.88 ± 0.38 (mean ± SD), the methylation of the LIPA promoter will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian Italian subjects
* age > 18 and < 70 years
* non-cirrhotic NAFLD

Exclusion Criteria:

* any malignant disease during the last 5 years
* any inflammatory or autoimmune disease
* corticosteroids for systemic use
* any medication potentially affecting body weight or body composition
* syndromic obesity
* renal failure (GFR<90 ml/min)
* heart failure (NYHA classes II-IV)
* any type liver disease rather than NAFLD
* alcohol intake >140g/ week for men and 70g/ week for women
* participation in a reducing- weight program in the last 3 months
* cholestyramine during the last 6 months before enrollment
* previous cholecystectomy
* gallbladder disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-cirrhotic NALFD patients, wild type for the PNPLA3 risk variant and with a LAL value in DBS of 0.88±0.38 (mean±SD) and non-cirrhotic NALFD patients, carriers for PNPLA3 risk variant (heterozygous and mutant homozygous both) with a LAL value in DBS of 0.76±0.38 (mean±SD)
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Inhibition enzyme assay to test LAL activity | enrollment
  Activity of LAL enzyme will be measured in 158 subjects affected by non-cirrhotic NAFLD and wild type for the PNPLA3 rs738409 risk variant, in whole blood, plasma and platelets.
Inhibition enzyme assay to test LAL activity | enrollment
  Activity of LAL enzyme will be measured in 158 subjects affected by non-cirrhotic NAFLD and carriers for the PNPLA3 rs738409 risk variant, in whole blood, plasma and platelets.

SECONDARY OUTCOMES:
Inhibition enzyme assay to test LAL activity variation | 18 months
  Activity of LAL enzyme will be measured at 18 months respect to enrollment, in 158 subjects affected by non-cirrhotic NAFLD and wild type for the PNPLA3 rs738409 risk variant, in whole blood, plasma and platelets.
Inhibition enzyme assay to test LAL activity variation | 18 months
  Activity of LAL enzyme will be measured at 18 months respect to enrollment, in 158 subjects affected by non-cirrhotic NAFLD and carriers for the PNPLA3 rs738409 risk variant, in whole blood, plasma and platelets.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Translational and Precision Medicine, Sapienza University of Rome, Umberto I Hospital, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No